CLINICAL TRIAL: NCT06600997
Title: Parent Artery Reconstruction for Small Unruptured Cerebral Aneurusms Using Flow DiverTers: a Multicenter Randomized Trial(PARAT-MT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PARAT-MT
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Aneurysm Unruptured; Cerebral Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Flow diversion for endovascular treatment of intracranial aneurysms
  Interventions: Device: Flow Diversion for Endovascular Treatment of Intracranial Aneurysms
- Control group (Active Comparator): Conventional endovascular therapy (stent-assisted coiling, balloon-assisted coiling, or coiling) for endovascular treatment of intracranial aneurysms
  Interventions: Device: Conventional endovascular therapy (stent-assisted coiling, balloon-assisted coiling, or coiling) for endovascular treatment of intracranial aneurysms

INTERVENTIONS:
Device: Flow Diversion for Endovascular Treatment of Intracranial Aneurysms — Flow Diversion for Endovascular Treatment of Intracranial Aneurysms
  Arms: Intervention group
Device: Conventional endovascular therapy (stent-assisted coiling, balloon-assisted coiling, or coiling) for endovascular treatment of intracranial aneurysms — Conventional endovascular therapy (stent-assisted coiling, balloon-assisted coiling, or coiling) for endovascular treatment of intracranial aneurysms
  Arms: Control group

SUMMARY:
A prospective, multicenter, randomized controlled clinical trial with open-label treatment and blinded endpoint assessment.

DETAILED DESCRIPTION:
The PARAT-MT is to evaluate whether small unruptured cerebral aneurusm patients treated with FD superior to those treated with conventional endovascular therapy. It is a prospective, multicenter, randomized controlled clinical trial with open-label treatment and blinded endpoint assessment trial.

Primary Outcome Endpoint A composite endpoint of major recurrence, any stroke or death at one year post-surgery.

Second Outcome Endpoint

1. All-cause mortality at 12 months post-surgery.
2. Any stroke at 12 months post-surgery.
3. Major recurrence rate at 12 months post-surgery.
4. Transient ischemic attack (TIA) occurrence rate at 12 months post-surgery.
5. Periprocedural (30-day) procedure-related complications rate.
6. Ipsilateral stroke or neurologic death at 1 month and 12 months post-surgery
7. Severe disability rate at 1 month and 12 months post-surgery (mRS > 2).
8. Complete aneurysm occlusion rate at 12 months post-surgery (Raymond I).
9. The rate of in-stent stenosis ≥50% at 12 months post-surgery.
10. Incidence of hemorrhagic stroke at 12 months post-surgery.
11. Technical success rate.
12. Target parent artery retreatment rate at 12 months post-surgery.
13. Target aneurysm retreatment rate at 12 months post-surgery.
14. Surgical operation time.
15. Radiation dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Previously unruptured saccular cerebral aneurysm arising from intradural segments of the internal carotid artery and intracranial segments of the vertebral artery.
3. Measuring ≤10mm in maximum diameter
4. Subjects capable of understanding the study's purpose, willing to participate, and have signed an informed consent form.

Exclusion Criteria:

1. Subjects with two or more multiple aneurysms requiring treatment within one year.
2. Subjects with arteriovenous malformations or moyamoya disease.
3. Subjects with ruptured, recurrent, or dissecting aneurysms.
4. Subjects with symptomatic cerebral stenosis >70%;
5. Subjects who have experienced a stroke (cerebral hemorrhage, cerebral infarction) within the past month.
6. Clinical condition is extremely poor with a modified Rankin score of ≥3.
7. Subjects planned for surgical/interventional procedures within three months.
8. Subjects deemed inappropriate for interventional treatment by the investigator (e.g., no suitable vascular access, excessively tortuous vessels, difficult stent delivery, etc.).
9. Subjects with severe comorbidities, unsuitable for anesthesia or endovascular surgery (e.g., major cardiac, pulmonary, hepatic, splenic, renal diseases, atrial fibrillation ,brain tumors, severe active infections, disseminated intravascular coagulation, history of severe mental illness).
10. Subjects unable to tolerate antiplatelet or anticoagulant therapy.
11. Subjects who has had or are likely to have a severe reaction to contrast media.
12. Subjects with a history of allergy to nickel-titanium, cobalt-chromium, or platinum-tungsten alloys.
13. Subjects who have participated in other drug or medical device clinical trials and have not reached the primary endpoint time limit.
14. Pregnant or breastfeeding women.
15. Subjects with an expected lifespan of less than 12 months.
16. Subjects deemed by the investigator to have poor compliance, unable to complete the study as required.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1008 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2031-10-30 (Estimated)

PRIMARY OUTCOMES:
Major recurrence, any stroke or death | At 1 year post-surgery
  A composite endpoint of major recurrence, any stroke or death

SECONDARY OUTCOMES:
All-cause mortality | At 12 months post-surgery
  All-cause mortality
Any stroke | At 12 months post-surgery
  Any stroke
Major recurrence | At 12 months post-surgery
  Major recurrence
Transient ischemic attack (TIA) | At 12 months post-surgery
  Transient ischemic attack (TIA)
Procedure-related complications | Periprocedural (30 days)
  Procedure-related complications
Ipsilateral stroke or neurologic death | At 1 month and 12 months post-surgery
  Ipsilateral stroke or neurologic death
Severe disability | At 1 month and 12 months post-surgery
  Severe disability (mRS > 2)
Complete aneurysm occlusion | at 12 months post-surgery
  Complete aneurysm occlusion (Raymond I)
The rate of in-stent stenosis ≥50% | At 12 months post-surgery
  The rate of in-stent stenosis ≥50%
hemorrhagic stroke | at 12 months post-surgery
  Incidence of hemorrhagic stroke
Technical success rate | 24 hours after endovascular treatment
  Technical success rate
Target parent artery retreatment rate | At 12 months post-surgery
  Target parent artery retreatment rate
Target aneurysm retreatment rate | At 12 months post-surgery
  Target aneurysm retreatment rate
Surgical operation time | during surgery
  Surgical operation time
Radiation dose | during surgery
  Radiation dose

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, MD, PhD, Principal Investigator — Changhai Hospital

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with bona fide researchers after the publication of the main results, based on a submitted protocol to Oriental Collaboration group on Emerging Advanced therapy for Neurovascular diseases Consortium.
Supporting Information: Study Protocol, SAP
Time Frame: Data sharing will be available from 12 months after the publication of the main results.
Access Criteria: 1. The data sharing will be only for the purposes of health and medical research and within the constraints of the consent under which the data were originally gathered.
  2. The Custodian of the Collection will not consider any Proposals for data sharing that unblind, or potentially unblind, randomised comparisons in active / ongoing trials.
  3. Requesters should be employees of a recognised academic institution, health service organisation, commercial research organisation or from the pharmaceutical industry. Requesters must have experience in medical research.
  4. Requesters must be able to demonstrate through their peer review publications in the area of interest their ability to carry out the proposed use of the requested dataset from a Collection.
  5. The Requesters must not have a conflict of interest that may potentially influence their interpretation of any analyses.
URL: https://www.ocin.org.cn/